CLINICAL TRIAL: NCT00740480
Title: A Prospective, Non-Randomized, Limited-Use Evaluation of the ENTact Septal Staple System for Tissue Approximation During Septoplasties
Brief Title: Study of the ENTact Septal Staple System for Tissue Approximation During Septoplasty
Status: Completed | Type: Observational
Sponsor: ENTrigue Surgical, Inc. (Industry)
Responsible Party: Gabriele Niederauer, Ph.D./Vice President, Research and Development, ENTrigue Surgical, Inc.
Other Study IDs: CSA 2008-01
Record Dates: First submitted 2008-08-21; First posted 2008-08-25 (Estimated); Results first posted 2009-08-21 (Estimated); Last update posted 2009-08-25 (Estimated); Status verified 2009-08

CONDITIONS: Nasal Septum
Keywords: Evaluation; ENTact™; Septal; Staple; System; tissue; approximation; during; septoplasties

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Surgical: Adult population (ages 18-65) with clinically significant nasal septum deviation.

SUMMARY:
The purpose of this research study is to learn more about the ENTact™ Septal Staple System device performance and to collect information to support its premarket application.

DETAILED DESCRIPTION:
The ENTact™ Staple System is a device that inserts a small staple or tack to hold mucosa (moist tissues) in place instead of using stitches. The staple gradually dissolves and does not need to be removed. This clinical study will evaluate:

* surgical performance of the ENTact Septal Staple System
* one week post op clinical evaluation of gross tissue appearance at implantation site(s)
* ENTact™ Septal Staple functionality based on maintained coaptation

ELIGIBILITY:
Inclusion Criteria:

* Adult patients, between the ages of 18 and 65 years, with a clinically significant deviation of the nasal septum
* Patient is able to provide a signed informed consent form
* Patient will agree to comply with all study related procedures
* Patient is not pregnant at this time. If patient is of child-bearing age and capable of bearing children, a pre-operative pregnancy test confirmation is required to show that patient is not pregnant on the day of surgery
* Patient does not plan on becoming pregnant and is not breast feeding during the course of the study

Exclusion Criteria:

* Patients who do not meet the inclusion criteria
* Patients who have had previous septoplasty
* Patients with uncontrolled diabetes
* Presence of infection at the site
* Smokers and severe drug and alcohol abusers
* Patients with autoimmune disease deemed clinically significant by Principal Investigator

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adult patients (ages 18-65) with clinically significant nasal septum deviation.
Sampling Method: Non-Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2008-04; Primary Completion 2009-02 (Actual); Study Completion 2009-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gabriele G Niederauer, Ph.D., Study Director — ENTrigue Surgical, Inc.
Locations (3):
- United States (3):
  - Good Samaritan Hospital, Cincinnati, Ohio
  - Park Hudson Surgery Center, Bryan, Texas
  - Physician's Ambulatory Surgery Center IV, San Antonio, Texas

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Chart reviews and patient contact in clinic. Recruitment period from July 2008 to January 2009.
Groups:
- Septal Stapler Group: Adult population (ages 18-65) with clinically significant nasal septum deviation.
Period: Overall Study
Arm/Group | Septal Stapler Group
Started | 25
Completed | 23
Not Completed | 2
Not completed — Adverse Event | 1
Not completed — Physician Decision | 1

BASELINE CHARACTERISTICS:
Arm/Group | Septal Stapler Group
Number analyzed (Participants) | 25
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 25
  >=65 years | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 39.9 (13.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 12
Region of Enrollment [Number; unit: participants]
  United States | 25

OUTCOME MEASURES:

1. Primary Outcome: Coaptation (Tissue Approximation)
Description: Complete tissue approximation at one week.
Time Frame: One week post surgery
Population: ITT
Measure: Number; unit: participants
Arm/Group | Septal Stapler Group
Number analyzed (Participants) | 25
participants | 23

2. Secondary Outcome: Tissue Reaction to Implant
Description: None - no edema, erythema or purulence around the area of the staples Mild - slight erythema and/or edema in the region of one or more staple, limited to not greater than 2 mm from the staple Moderate - erythema and/or edema in the region of one or more staples, greater than 2 mm extension from the staples Severe - Generalized edema and/or erythema of the septum, or purulence and/or granulation tissue involved in one or more staples.
Time Frame: One week post surgery
Population: ITT
Measure: Number; unit: participants
Arm/Group | Septal Stapler Group
Number analyzed (Participants) | 25
participants
  No reaction | 18
  Mild reaction | 5
  Moderate reaction | 0
  Severe reaction | 0
  Cannot assess | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No